CLINICAL TRIAL: NCT01201044
Title: A Randomized, Two Arm Study to Investigate Bronchial Arterrial Infusing (BAI) Plus Three-dimensional Conformal Radiotherapy (3DCRT) in Local Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: Study to Investigate Bronchial Arterrial Infusing (BAI) Plus Three-dimensional Conformal Radiotherapy (3DCRT) in Local Advanced Non-small Cell Lung Cancer (NSCLC)
Acronym: DO201001
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Yi Li, The Third Affiliated of the The Third Military Medical University Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DO201001; DO210101
Record Dates: First submitted 2010-05-24; First posted 2010-09-14 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2009-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: BAI; 3DCRT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; nedaplatin; Bays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemcitabine, Nedaplatin,BAI plus 3DCRT (Experimental): Gemcitabine(1000mg/m2)，Nedaplatin(60mg/m2),BAI, Day 1/4weeks. 4weeks per cycle. Tumor assessment will be perforemd after 2 cycles. if no PD, patient will be treated with 3DCRTfor 1 month. for patient PD after 3DCRT, complete the study. patient no PD after 3DCRT will receive 2 cycle of chemo with Gemcitabine. Nedaplatin.
  then patient will be followed for 1 year..
  Interventions: Radiation: 3DCRT; Drug: Gemcitabine，Nedaplatin, BAI
- Gemcitabine, Nedaplatin, IV Plus 3DCRT (Other): Gemcitabine 100mg/m2, D1 & D8 every 4 weeks Nedaplatin 75mg/m2, D1 every 4 weeks. every 4 weeks per cycle. Tumor assessment will be performed after 2 cycles. if no PD, patient will be treated with 3DCRT for 1 month.
  for patient PD after 3DCRT, complete the study. patient no PD after 3DCRT will receive 2 cycle of chemo with Gemcitabine. Nedaplatin.
  then patient will be followed for 1 year.
  Interventions: Drug: Gemcitabine, Nedaplatin, iV; Radiation: 3DCRT

INTERVENTIONS:
Drug: Gemcitabine, Nedaplatin, iV — Gemcitabine, Injection, 1000mg/m2, D1 & D7/ 4weeks/cycle, 2 cycles Nedaplatin, Injection, 75mg/m2, d1/4weeks/cycle, 2 cycles.
  Arms: Gemcitabine, Nedaplatin, IV Plus 3DCRT
Radiation: 3DCRT — non-PD Patient will be treated with 3DCRT after 2 cycles of chemo.
  Arms: Gemcitabine, Nedaplatin, IV Plus 3DCRT
Radiation: 3DCRT — non-PD Patient will be treated with 3DCRT after 2 cycles of chemo.
  Arms: Gemcitabine, Nedaplatin,BAI plus 3DCRT
Drug: Gemcitabine，Nedaplatin, BAI — Drug: Gemcitabine, Nedaplatin, iV
  Gemcitabine, Injection, 1000mg/m2, D1/4weeks/cycle, 2 cycles Nedaplatin, Injection, 75mg/m2, d1/4weeks/cycle, 2 cycles. BAI
  Arms: Gemcitabine, Nedaplatin,BAI plus 3DCRT

SUMMARY:
The purpose of this study is to investigate the efficacy of BAI Plus 3DCRT in local advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* stage IIIA&IIIB NSCLC
* male or female, Age ≥18Years, ≤70Years
* Life expectation of at least 12weeks.
* PS performance 0-2
* Measurable disease according to the Response Evaluation Criteria in Solid Tumours ( RECIST)

Exclusion Criteria:

* Patient with prior chemotherapy or radiology for IIIA or IIIB NSCLC

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | every 2 cycles
  Regular tumour assessments (based on RECIST criteria) for determining disease response and progression using CT and MRI scans, and overall survival.The primary efficacy variable is progression free survival (PFS), defined as the time between randomisation and the date of first documented disease progression or death from any cause, whichever comes first. Disease progression is defined according to the RECIST criteria.

SECONDARY OUTCOMES:
Overall Survival | every 3 month after Progressive Disease
  after Progressive Disease, patient will be contact every 3 month for the survival information.
Time to Progressive Disease (RECIST Criteria) | Every 2 cycles
  Regular tumour assessments (based on RECIST criteria) for determining disease response and progression using CT and MRI scans.Time to Progression (TTP) is defined as the time between randomisation and the date of the first documented disease progression.

CONTACTS AND LOCATIONS:
Locations (1):
- The 3rd Affiliated Hospital of the 3rd Military Hospital, Chongqing, China